CLINICAL TRIAL: NCT05476627
Title: Risk Factors and Multiomics Study of Chronic Kidney Disease Caused by Metabolic Diseases
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Limeng Chen, director of the department of nephrology, Peking Union Medical College Hospital
Other Study IDs: JS-2136
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Chronic Kidney Diseases; Hypertension; Diabetes Mellitus; Hyperuricemia; Obesity
Keywords: chronic kidney disease; metabolic diseases; biomarker; functional imaging techniques
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension; Diabetes Mellitus; Hyperuricemia; Obesity; Metabolic Diseases | interventions — Environmental Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Hypertension Group
  Interventions: Diagnostic Test: Biomarkers
- Diabetes Group
  Interventions: Diagnostic Test: Biomarkers
- Hyperuricemia
  Interventions: Diagnostic Test: Biomarkers
- Obesity
  Interventions: Diagnostic Test: Biomarkers

INTERVENTIONS:
Diagnostic Test: Biomarkers — Blood,urine and imaging biomarkers for early diagnosis and prediction of prognosis.

SUMMARY:
With the development of China's economy, people's living standard have improved, and the dietary structure have changed. Metabolic diseases, such as hypertension, diabetes, hyperuricemia and obesity have gradually become an important health burden in China. The pathophysiological mechanism of renal injury caused by metabolic diseases has always been a hotspot of research. Currently, it is believed that various mechanisms including the activation of Renin-Angiotensin-Aldosterone System, vascular endothelial dysfunction, oxidative stress and inflammatory process may be involved. Although there are differences in renal pathological manifestations caused by different metabolic diseases, the kidney will eventually present ischemic changes and fibrosis with the progression of the disease. So there must be some common pathogenesis. This study is designed to build a disease cohort of patients with chronic kidney disease caused by metabolic diseases, to identify risk factors leading to disease progression and to explore biomarkers for early diagnosis and treatment of kidney damage.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of metabolic diseases were confirmed;
* Be able to understand the process of the research;
* Volunteer for participation and be able to sign the informed consent.

Exclusion Criteria:

* Age <18 yrs or >80yrs;
* Patients with primary and secondary glomerular diseases
* Patients with other comorbidities that could affect the volume or the components of the kidney, such as renal cysts, polycystic kidney disease, medullary sponge kidney, hydronephrosis, renal artery stenosis, renal vein thrombosis and/or renal tumors;
* Contraindications for MRI examination;
* Pregnant or lactation patients;
* Patients with unstable vital signs, failure of other organs or dysphoria.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is consecutively enrolled from outpatient and inpatient department of our hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with End Stage Renal Disease | 3 years
  End Stage Renal Disease
Number of Participants with Adverse cardiovascular events | 3 years
  Adverse cardiovascular events
Number of Participants with all cause death | 3 years
  All cause death

SECONDARY OUTCOMES:
Number of Participants with eGFR decline | 3 years
  the decline of eGFR during follow-up
Number of Participants with Complications of CKD | 3 years
  The complications of CKD
Life quality assessment with short form-36 (SF-36) | 3 years
  The SF-36 is a patient-reported instrument designed to assess overall health status; it is usually utilized to measure patients' quality of life and used primarily in research. Increasing SF-36 scores are indicative of improving health status.
Advanced Intelligence Assessment with Mini-Mental State Examination (MMSE) | 3 years
  The MMSE is scored on a 30-point scale, with items that assess orientation (temporal and spatial; 10 points), memory (registration and recall; 6 points), attention/concentration (5 points), language (verbal and written; 8 points), and visuospatial function (1 point) . While different cutoff points have been used across studies, scores ≤23 are most commonly regarded as abnormal and indicative of cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Limeng Chen, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
De-privatized data are to be shared with other researchers.